CLINICAL TRIAL: NCT02297737
Title: Developing a Mindfulness Movement Intervention Program for Post-MI Patients: A Randomized 75-subject Pilot Clinical Trial of Tai Chi Versus Health Education in Post-myocardial Infarction Patients
Brief Title: Mindful Movement Intervention for Post-MI Patients
Acronym: HeartChi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura S. Redwine, PhD, Asst Adjunct Prof, San Diego Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1R21AT007600-01A1 (NIH)
Record Dates: First submitted 2014-09-19; First posted 2014-11-21 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Myocardial Infarction
Keywords: Tai Chi
MeSH Terms: conditions — Myocardial Infarction | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi (Experimental): A manual consisting of 8 movements learned over a period of 12 weeks will be used to teach participants in the Tai Chi condition. Classes will include around 5-6 subjects, each class lasting one hour, including a 10-minute warm-up and cool-down, and meet twice per week. Patients will be told to practice Tai Chi three times/week at home. After 12 weeks of training patients will be told to practice at home five times/week for 8 more weeks, until the 8-week follow-up visit. Subjects will be asked to rate their perceived exertion/work intensity during each session using the Borg's perceived exertion scale and asked to increase the size of their movements to reach 12-13 (moderate difficulty), which consistently matches with 65-70% of HR max.
  Interventions: Behavioral: Tai Chi
- Health Education (Active Comparator): Participants in the Health Education condition will also meet for one hour, twice per week for 12 weeks for a total of 24 hours. Sessions will be highly structured and will emphasize key concepts in the presentations. Medical and allied health experts will provide twelve didactic videotaped presentations on a series of health-related themes and a group leader will be present to answer questions. Themes will include: Epidemiology of Cardiovascular Disease, Patient/Physician Communication, Medication Adherence, Nutrition and Exercise, The Nature and Structure of Sleep, and Navigating the Health Care System.
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: Tai Chi
  Arms: Tai Chi
Other: Health Education
  Arms: Health Education

SUMMARY:
This study evaluates the feasibility and acceptability of a 12-week Tai Chi intervention for patients who have recently had a heart attack and are not participating in a standard cardiac rehabilitation program. Half of the 75 patients will be randomly assigned to the Tai Chi condition and the other half will be assigned to 12 weeks of Health Education. In addition to examining feasibility and acceptability, the investigators will evaluate the impact of participation in the Tai Chi condition on measures of cardiac health, physical function, self-reported health behaviors, and mental health as compared to Health Education within the context of this developmental/exploratory study.

DETAILED DESCRIPTION:
Each year around 785,000 Americans endure a first heart attack and more than half will have another in the future. The American Heart Association (AHA) recommends exercise-based cardiac rehabilitation (CR) to aid prevention of future heart attacks. Despite the benefits of CR, only a small proportion of eligible patients participate in CR. Patients with other illnesses, women, older adults, and ethnic minorities are least likely to utilize CR services. Many medical centers do not have CR programs and patients have to travel to distant locations to undergo CR. In turn, Tai Chi has been studied in the elderly, requires no expensive equipment, can be practiced at home, and is well tolerated across fitness levels and co-occurring illnesses. Tai Chi serves as an aerobic exercise of low to moderate intensity. However, no Tai Chi studies in post-MI patients have employed state-of-the-art measures of cardiac function and exercise capacity and therefore it is unclear whether Tai Chi has similar benefits as CR during the period of recovery from a heart attack. This study is innovative in that it specifically targets patients who have not opted to participate in a formal CR program within 6 months of a first-time heart attack and emphasizes recruitment of patients spanning an older age range, physical function ability, women and minorities. A total of 75 men and women with a first time heart attack will be randomly assigned to 24 sessions of Tai Chi training composed of 8 meditative movements or to an equivalent "dose" of Health Education classes. Clinical assessments will be performed over a 4-5 month period, with testing occurring before, mid-way, after treatment, and at an 8-week follow-up. Our goal is to gather preliminary data on study feasibility, acceptability and to find indications of improvements in measures of cardiac health, physical function, health behaviors, and mental health. If the aims are met from this exploratory/development study, a future large scale study will be undertaken to confirm Tai Chi's effectiveness in post-heart attack patients. Such research is critically needed to aid the development of effective rehabilitative interventions that will be acceptable to a wider range of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Suffered an MI (ST Elevation MI (STEMI) or Non-ST Elevation MI (NSTEMI) with creatine kinase MB fraction elevation 3 times the upper limits of normal and with ischemic ECG changes within 6 months of baseline testing;
2. Clinically stable---defined as no active arrhythmia, no residual ischemia;
3. Able to perform light to moderate exercise;
4. Able to give informed consent, understand study procedures and to comply with them for the entire length of the study;
5. A 30 day period since Percutaneous Coronary Intervention (PCI);
6. Medical clearance by their cardiologist;
7. "Treatment as usual" medications prescribed by their cardiologist (see allowed medications under 6.2. Description of Evaluations);
8. Antidepressant treatment with SSRIs or SNRIs is allowed, but not required;
9. > 35 years of age.

Exclusion Criteria:

1. Unstable angina;
2. Severe valvular disease;
3. Severe COPD;
4. Recent stroke or significant cerebral neurologic impairment;
5. Moderate to severe suicidal risk (BDI-II #9 > 1 or from the SCID interview for MDD);
6. Cancer;
7. Currently in an exercise program;
8. Current uses of mood stabilizers, or antipsychotics;
9. Medications (steroids) and conditions affecting immune status
10. Pregnant, lactating or intending to become pregnant;
11. Meets criteria for bipolar disorder, schizophrenia, substance use disorder
12. Currently taking benzodiazepines and mood stabilizers
13. Inability to give written informed consent in English.
14. Participation in another intervention study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility, Treatment Expectancy/Satisfaction, Retention, and Adherence (Recruitment rates) | Two years
  Recruitment rates will be recorded.
Feasibility, Treatment Expectancy/Satisfaction, Retention, and Adherence (Barriers to CR) | Two years
  Barriers to CR will be queried at baseline and at the end of the interventions to determine changes in attitudes.
Feasibility, Treatment Expectancy/Satisfaction, Retention, and Adherence (6-item credibility/expectancy questionnaire (CEQ) | Two years
  A 6-item credibility/expectancy questionnaire (CEQ) will be measured at baseline and monthly to determine Tai Chi and Health Education acceptability.
Feasibility, Treatment Expectancy/Satisfaction, Retention, and Adherence (retention rates, exit interviews) | Two years
  Retention rates will be recorded, and exit interviews administered to determine reasons for drop-out. Adherence to exercise in general, and Tai Chi specifically, will be derived from exercise logs. The Exercise Benefits/Barriers Scale (EBBS) will be administered at baseline and each time point and an exit interview on the post-intervention visit will query barriers to attending Tai Chi classes and practice, as well as attendance of Health Education classes.

SECONDARY OUTCOMES:
Physical function (Six-minute walk test) | Five months
  Six-minute walk test
Psychological and health behaviors (Beck Depression Inventory) | Five months
  Beck Depression Inventory
Biomarkers of cardiac risk (CRP, BNP, sST2) | Five months
  Inflammatory Biomarkers (CRP, BNP, sST2)
Cardiac Function (Blood pressure and heart rate) | Five months
  Blood pressure and heart rate
Psychological and health behaviors (Cardiac Self-Efficacy Questionnaire) | Five Months
  Cardiac Self-Efficacy Questionnaire
Psychological and health behaviors (Five Facets of Mindfulness Questionnaire) | Five Months
  Five Facets of Mindfulness Questionnaire
Psychological and health behaviors (Functional Assessment of Chronic Illness Therapy--Spiritual Well-Being Scale) | Five Months
  Functional Assessment of Chronic Illness Therapy--Spiritual Well-Being Scale
Psychological and health behaviors (Goldberg Anxiety and Depression Scale) | Five Months
  Goldberg Anxiety and Depression Scale
Psychological and health behaviors (Morisky 8-item Medication Adherence Scale) | Five Months
  Morisky 8-item Medication Adherence Scale
Psychological and health behaviors (Perceived Stress Scale) | Five Months
  Perceived Stress Scale
Psychological and health behaviors (Pittsburgh Sleep Quality Index) | Five Months
  Pittsburgh Sleep Quality Index
Psychological and health behaviors (Positive and Negative Affect Schedule) | Five Months
  Positive and Negative Affect Schedule
Psychological and health behaviors (Short Form--12 Health Survey) | Five Months
  Short Form--12 Health Survey
Psychological and health behaviors (SCID-I N/P Mood Module) | Five Months
  SCID-I N/P Mood Module,

CONTACTS AND LOCATIONS:
Overall Officials: Laura S Redwine, PhD, Principal Investigator — University of California, San Diego